CLINICAL TRIAL: NCT00460200
Title: Depression and IL-6 in Epithelial Ovarian Cancer: Genetic Diathesis and Psychological Stress
Brief Title: Depression and Interleukin-6 Production in Patients With Ovarian Epithelial Cancer
Status: Withdrawn | Type: Observational
Why Stopped: no patient accrual
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000385692; UCLA-0309083-01; UCLA-002
Record Dates: First submitted 2007-04-11; First posted 2007-04-13 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-10

CONDITIONS: Depression; Fatigue; Ovarian Cancer; Psychosocial Effects of Cancer and Its Treatment; Sleep Disorders
Keywords: depression; fatigue; sleep disorders; psychosocial effects of cancer and its treatment; ovarian epithelial cancer
MeSH Terms: conditions — Depression; Fatigue; Ovarian Neoplasms; Sleep Wake Disorders; Carcinoma, Ovarian Epithelial | interventions — Amplified Fragment Length Polymorphism Analysis; Therapeutics; Psychiatric Rehabilitation

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: polymorphism analysis
Other: laboratory biomarker analysis
Other: physiologic testing
Other: questionnaire administration
Procedure: conventional surgery
Procedure: fatigue assessment and management
Procedure: psychosocial assessment and care

SUMMARY:
RATIONALE: Measuring levels of interleukin-6 and depression may help doctors understand the relationship between interleukin-6 and depression. It may also help the study of cancer in the future.

PURPOSE: This clinical trial is studying depression and interleukin-6 production in patients with ovarian epithelial cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Correlate tumor production of interleukin (IL)-6, serum levels of IL-6, and IL-6 coding or promoter single nucleotide polymorphisms with IL-6 protein production in patients with ovarian epithelial cancer.
* Correlate tumor culture supernatant, ascitic fluid, and/or serum IL-6 level with levels of depression and/or anxiety in these patients to determine whether catecholamines or cortisol may alter production of IL-6 by cultured ovarian cancer cells.
* Determine the effects of neuroendocrine activity on modulation of IL-6 production in these patients.
* Compare immune response to autologous tumor tissue in "MLR-like" reactions between tumor and peripheral blood mononuclear cells in vitro.
* Correlate the levels of immunologic response with relapse and/or survival times, clinical response to CA 125 antibody treatment (e.g., in a pre- vs post-therapy sampling framework), and IL-6 parameters in these patients.
* Determine the use of epitope prediction bioinformatic tools in consultation with Coulter to set up a major histocompatibility complex (MHC) tetramer assay for assessing cytotoxic T lymphocyte levels in peripheral blood from these patients.
* Determine the incidence of herpes virus infections in these patients.

OUTLINE: This is a pilot study.

Before and after cytoreduction surgery, patients complete multiple questionnaires, including Beck Depression Inventory, Positive & Negative Mood State, Fatigue Symptom Inventory, Revised NEO Personality Inventory, COPE, SF-36, Pittsburgh Sleep Quality Inventory, and Mental Adjustment to Cancer, to assess depression and coping mechanisms.

Blood samples are collected at baseline and on postoperative days 1-4 and analyzed for interleukin (IL)-6, c-reactive protein, herpes simplex virus-8 (HSV8), epinephrine, adrenocorticotropic hormones, and cortisol. Ovarian carcinoma tissue samples and peritoneal fluid are also collected and evaluated for production and utilization of IL-6, HSV8, and autonomic nervous system and hypothalamic-pituitary-adrenal activity.

PROJECTED ACCRUAL: Approximately 36 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of ovarian epithelial cancer
* Scheduled to undergo cytoreduction of ovarian tumor

PATIENT CHARACTERISTICS:

* Able to communicate with the investigator

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: diagnosis of ovarian epithelial cancer
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2003-12

PRIMARY OUTCOMES:
Correlation of tumor production of interleukin (IL)-6, serum levels of IL-6, and IL-6 coding or promoter single nucleotide polymorphisms with IL-6 protein production
Correlation of tumor culture supernatant, ascitic fluid, and/or serum IL-6 level with levels of depression and/or anxiety
Effects of neuroendocrine activity on modulation of IL-6 production
Comparison of immune response to autologous tumor tissue in "MLR-like" reactions between tumor and peripheral blood mononuclear cells in vitro
Correlation of levels of immunologic response with relapse and/or survival times, clinical response to CA 125 antibody treatment, and IL-6 parameters
Establishment of a major histocompatibility complex (MHC) tetramer assay for assessing cytotoxic T lymphocyte levels in peripheral blood
Incidence of herpes virus infections

CONTACTS AND LOCATIONS:
Overall Officials: Leah Z. Fitzgerald, RN, PhD, Principal Investigator — Jonsson Comprehensive Cancer Center